CLINICAL TRIAL: NCT05325866
Title: A Phase 1b/2, Multicenter, Open-label Basket Study Evaluating the Safety and Efficacy of Bemarituzumab Monotherapy in Solid Tumors With FGFR2b Overexpression (FORTITUDE-301)
Brief Title: A Study Evaluating Bemarituzumab in Solid Tumors With Fibroblast Growth Factor Receptor 2b (FGFR2b) Overexpression
Acronym: FORTITUDE-301
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20210104; 2023-505455-44 (EudraCT Number)
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors
Keywords: Epithelial solid tumors with fibroblast growth factor receptor 2b overexpression; FGFR2b; Head and neck squamous cell carcinoma; Triple-negative breast cancer; Intrahepatic cholangiocarcinoma; Lung adenocarcinoma; Ovarian epithelial carcinoma; Endometrial adenocarcinoma; Cervical carcinoma; Bemarituzumab; AMG 552; Other solid tumors
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms; Cholangiocarcinoma; Adenocarcinoma of Lung; Carcinoma, Ovarian Epithelial; Uterine Cervical Neoplasms | interventions — bemarituzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Monotherapy Dose Exploration (Experimental): Participants across multiple primary epithelial solid tumors with centrally determined FGFR2b overexpression and relapsed/refractory unresectable and/or metastatic disease will receive 1 of 2 dose regimens of bemarituzumab to determine recommended Phase 2 dose.
  Interventions: Drug: Bemarituzumab
- Part 2: Monotherapy Dose Expansion (Experimental): Participants across multiple primary epithelial solid tumors with centrally determined FGFR2b overexpression and relapsed/refractory unresectable and/or metastatic disease will receive the dose of bemarituzumab identified as the recommended Phase 2 dose during Part 1.
  Interventions: Drug: Bemarituzumab

INTERVENTIONS:
Drug: Bemarituzumab — Intravenous (IV) infusion.
  Other Names: AMG 552

SUMMARY:
The primary objectives of this study are to observe the safety and tolerability of bemarituzumab and to evaluate preliminary antitumor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years (or legal adult age within country, whichever is older) at the time that the Informed Consent Form (ICF) is signed
2. Histologically or cytologically confirmed cancer of one of the following types, refractory to or relapsed after at least 1 prior standard therapeutic regimen in the advanced/metastatic setting, as specified below. If no standard of care therapies exist for the participant, or the participant cannot tolerate or refuses standard of care anticancer therapy, the participant may be allowed to participate on the study after discussion between the investigator and Amgen medical monitor. Participants who have not received all approved or standard treatments for their cancer must be informed that these alternatives to receiving bemarituzumab are available prior to consenting to participate in the trial.

   * head and neck squamous cell carcinoma: ≥ 1 line of therapy
   * triple-negative breast cancer: ≥ 2 lines of therapy
   * Intrahepatic cholangiocarcinoma ≥ 1 line of therapy
   * lung adenocarcinoma: at least platinum-based chemotherapy, checkpoint inhibitor, and targeted therapy
   * platinum resistant ovarian epithelial cell carcinoma, including fallopian tube cancers and primary peritoneal cancers, defined as progression during or within 6 months of a platinum containing regimen: ≥ 1 line of therapy
   * endometrial adenocarcinoma: ≥ 1 line of therapy
   * cervical carcinoma: ≥ 1 line of therapy
   * other solid tumors: ≥ 1 line of therapy
3. Disease that is unresectable, locally advanced, or metastatic (not amenable to curative therapy)
4. Tumor overexpresses FGFR2b as determined by centrally performed immunohistochemistry (IHC) testing
5. Measurable disease per Response Evaluation Criteria in Solid Tumors Version 1.1
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Adequate organ function as determined per protocol.

Exclusion Criteria:

1. Untreated or symptomatic central nervous system (CNS) metastases or leptomeningeal disease.
2. Other solid tumor cohort excludes primary tumors of the CNS, squamous non-small cell lung cancer, gastric adenocarcinoma, and gastroesophageal junction adenocarcinoma
3. Impaired cardiac function or clinically significant cardiac disease including: unstable angina within 6 months prior to first dose of study treatment, acute myocardial infarction ≥ 6 months prior to first dose of study treatment, New York Heart Association (NYHA) class II-IV congestive heart failure, uncontrolled hypertension (defined as an average systolic blood pressure ≥ 160 mmHg or diastolic ≥ 100 mmHg despite optimal treatment, uncontrolled cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin, active coronary artery disease or corrected QT interval QTc ≥ 470
4. History of systemic disease or ophthalmologic disorders requiring chronic use of ophthalmic steroids
5. Evidence of any ongoing ophthalmologic abnormalities or symptoms that are acute (within 4 weeks) or actively progressing
6. Unwillingness to avoid use of contact lenses during study treatment and for at least 100 days after the end of treatment
7. Recent (within 6 months) corneal surgery or ophthalmic laser treatment or recent (within 6 months) history of, or evidence of, corneal defects, corneal ulcerations, keratitis, or keratoconus, or other known abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer prior/concomitant therapy
8. Prior treatment with any investigational selective inhibitor of the fibroblast growth factor (FGF)/FGF receptor pathway (unless approved standard of care for tumor indication).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants Who Experience a Dose Limiting Toxicity (DLT) | Day 1 to Day 28
Part 1: Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE) | Day 1 to 28 days after last dose (a maximum of 2 years)
  Adverse events (AEs) are defined as any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurs after the participant has received study treatment. Any clinically significant changes in vital signs, visual acuity, and clinical laboratory tests that occur after study treatment administration will be recorded as TEAEs.
Part 1: Number of Participants Who Experience a Treatment-related Adverse Event | Day 1 to 28 days after last dose (a maximum of 2 years)
Part 2: Objective Response (OR) Rate | Up to approximately 2 years
  OR = complete response (CR) + partial response (PR), measured by computed tomography (CT) or magnetic resonance imaging (MRI) as determined by investigator per Response Evaluation Criteria in Solid Tumors (RECIST v1.1).

SECONDARY OUTCOMES:
Part 1: OR Rate | Up to approximately 2 years
  OR = CR + PR, measured by CT or MRI as determined by investigator per RECIST v1.1.
Parts 1 and 2: Disease Control (DC) Rate | Up to approximately 2 years
  DC = CR, PR, or stable disease (SD).
Parts 1 and 2: Duration of Response (DOR) | Up to approximately 2 years
  DOR, defined as the time from first documentation of OR (as determined by investigator per RECIST v1.1) until the first documentation of disease progression or death due to any cause, whichever occurs first. Only participants who have achieved OR will be evaluated for DOR. DOR will be censored at the last evaluable post-baseline tumor assessment prior to subsequent anticancer therapy.
Parts 1 and 2: Time to Response | Up to approximately 2 years
Parts 1 and 2: Progression-free Survival (PFS) | Up to approximately 2 years
  PFS, defined as time from first dose of investigational product until the first documentation of radiologic disease progression or death due to any cause. PFS will be censored at the last evaluable post-baseline tumor assessment prior to subsequent therapy. Progression will be based on RECIST v1.1 (derived utilizing investigator tumor assessments).
Parts 1 and 2: Overall Survival (OS) | Up to approximately 2 years
  OS, defined as time from first dose of investigational product until death from any cause. Participants still alive will be censored at the date last known to be alive.
Part 2: Number of Participants Who Experience a TEAE | Day 1 to 28 days after last dose (a maximum of 2 years)
  AEs are defined as any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are any event that occurs after the participant has received study treatment. Any clinically significant changes in vital signs, visual acuity, and clinical laboratory tests that occur after study treatment administration will be recorded as TEAEs.
Part 2: Number of Participants Who Experience a Treatment-related AE | Day 1 to 28 days after last dose (a maximum of 2 years)
Parts 1 and 2: Area Under the Concentration Time Curve (AUC) of Bemarituzumab | Day 1 to 28 days after last dose (a maximum of 2 years)
Parts 1 and 2: Maximum Observed Serum Concentration (Cmax) of Bemarituzumab | Day 1 to 28 days after last dose (a maximum of 2 years)
Parts 1 and 2: Observed Concentration at the End of a Dose Interval (Ctrough) of Bemarituzumab | Day 1 to 28 days after last dose (a maximum of 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (115):
- United States (10):
  - City of Hope National Medical Center, Duarte, California
  - University of California Irvine, Orange, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Community Health Network MD Anderson Cancer Center - North, Indianapolis, Indiana
  - Henry Ford Hospital, Detroit, Michigan
  - United States Oncology Regulatory Affairs Corporate Office, Nashville, Tennessee
  - Texas Oncology - Dallas Fort Worth, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - US Oncology Research Investigational Products Center, Irving, Texas
  - Texas Oncology Northeast Texas, Tyler, Texas
- Argentina (7):
  - Instituto Alexander Fleming, Capital Federal, Buenos Aires
  - Hospital Aleman, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fundacion Cenit Para La Investigacion, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Sociedad de Beneficencia Hospital Italiano, Córdoba, Córdoba Province
  - Fundacion Medica de Rio Negro y Neuquen, Cipolletti, Río Negro Province
  - Centro Oncologico Korben, Buenos Aires
- Australia (6):
  - Liverpool Hospital, Liverpool, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Toowoomba Hospital, Toowoomba, Queensland
  - Cabrini Hospital, Malvern, Victoria
  - St John of God Murdoch Hospital, Murdoch, Western Australia
- Austria (2):
  - Medizinische Universitaet Graz, Graz
  - Landeskrankenhaus Salzburg, Salzburg
- Belgium (5):
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Grand Hopital de Charleroi - Site des Viviers, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
- Brazil (7):
  - Hospital das Clinicas da Ufmg, Belo Horizonte, Minas Gerais
  - Centro de Oncologia Mackenzie, Curitiba, Paraná
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo, São Paulo
  - Beneficencia Portuguesa de Sao Paulo - Bp, São Paulo, São Paulo
  - Oncologia Rede D Or, São Paulo, São Paulo
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
- Bulgaria (3):
  - Multiprofile Hospital for Active Treatment Central Onco Hospital OOD, Plovdiv
  - Complex Oncology Center Plovdiv EOOD, Plovdiv
  - Military Medical Academy Multiprofile Hospital for Active Treatment - Sofia, Sofia
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- Rigshospitalet, København Ø, Denmark
- Finland (2):
  - Docrates Syopasairaala, Helsinki
  - Tampere University Hospital, Tampere
- France (8):
  - Institut de Cancerologie de l Ouest Rene Gauducheau, Angers
  - Centre Hospitalier Regional Universitaire de Besancon - Hopital Jean Minjoz, Besançon
  - Centre Oscar Lambret, Lille
  - Institut Paoli Calmettes, Marseille
  - Institut regional du Cancer Montpellier, Montpellier
  - Hopital Lyon sud, Pierre-Bénite
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Greece (5):
  - Sotiria General Hospital, Athens
  - Alexandra Hospital, Athens
  - Metropolitan General, Athens
  - University Hospital of Heraklion, Heraklion - Crete
  - European Interbalkan Medical Center, Thessaloniki
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz Nyiregyhazi Josa Andras Tagkorhaz, Nyíregyháza
  - Jasz-Nagykun-Szolnok Varmegyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah Ein-Kerem Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Istituto di Candiolo Fondazione del Piemonte per l Oncologia IRCCS, Candiolo to
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - Azienda Unita Locale Socio Sanitaria 3 Presidio Ospedaliero di Mirano, Mirano
  - Ospedale del Mare, Napoli
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Policlinico Umberto I, Roma
- Japan (5):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
- Mexico (5):
  - Investigacion Onco Farmacéutica S de RL de CV, La Paz, Baja California Sur
  - Centro de Infusion e Investigacion Oncologia de Saltillo, Saltillo, Coahuila
  - Health Pharma Professional Research SA de CV, Mexico City, Mexico City
  - Investigacion Biomedica para el Desarrollo de Farmacos, Mexico City, Mexico City
  - Christus Muguerza Clinica Vidriera, Monterrey, Nuevo León
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Radboud Universitair Medisch Centrum, Nijmegen
- Poland (5):
  - Pratia Mcm Krakow, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Ars Medical Spzoo, Piła
  - Mazowiecki Szpital Wojewodzki im Sw Jana Pawla II w Siedlcach spzoo, Siedlce
  - Centrum Medyczne Pratia Poznan, Skorzewo
- Portugal (3):
  - Unidade Local de Saude de Lisboa Ocidental, EPE - Hospital Sao Francisco Xavier, Lisbon
  - Hospital da Luz, SA, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
- Romania (4):
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Centrul de Oncologie Sf Nectarie SRL, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - SC Oncomed SRL, Timișoara
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Quironsalud Barcelona, Barcelona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital General Universitario Gregorio Maranon, Madrid
- Switzerland (2):
  - Kantonsspital Graubuenden, Chur
  - Hopitaux Universitaires de Geneve, Geneva
- United Kingdom (2):
  - Christie Hospital, Manchester
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2 ) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com